CLINICAL TRIAL: NCT04974840
Title: Effects of Thera-band Resisted Treadmill Training on Walking Ability in Chronic Stroke Patients
Brief Title: Thera-band Resisted Treadmill Training for Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sang-I Lin (Other)
Responsible Party: Sponsor-Investigator, Sang-I Lin, Professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-110-027
Record Dates: First submitted 2021-07-16; First posted 2021-07-23 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Chronic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill training combined with thera-band (Experimental): Participants will receive walking training on treadmill with thera-band at the waist. The direction of the thera-band resistance will be straight backward, backward-toward-right, and backward-toward-left. For each direction, the level of resistance and treadmill speed will be adjusted to allow the participants to perceive a 10-minute training to be 'slightly difficult'.
  Interventions: Behavioral: Treadmill training combined with/ without thera-band
- Treadmill training alone (Active Comparator): Participants will receive treadmill walking training at a speed that will be adjusted to allow the participants to perceive a 10-minute training to be 'slightly difficult'. For each session, there will be three 10-min treadmill walking bouts.
  Interventions: Behavioral: Treadmill training combined with/ without thera-band

INTERVENTIONS:
Behavioral: Treadmill training combined with/ without thera-band — Treadmill walking training with thera-band Treadmill walking training without thera-band

SUMMARY:
The purpose of this study is to determine if treadmill training combined with thera-band resistance to body support and forward propulsion would be more effective than treadmill training alone in improving over-ground walking ability and reducing energy cost in chronic stroke patients. This study will also characterize the neuromuscular and kinematic strategies to adapt to resisted treadmill walking in non-impaired adults and stroke patients.

DETAILED DESCRIPTION:
This study includes chronic stroke patients who will be randomly assigned to treadmill training combined with thera-band or treadmill training alone group to receive 30 min per session, 2 sessions per week for 8 weeks walking training . Functional balance (Berg Balance Scale), gait characteristics during preferred and maximal speed level walking, and oxygen uptake during 5-minute bouts of treadmill walking will be assessed before and after training and at 2-month follow-up. Clinical sensorimotor function assessment, including hand grip strength, plantar sensitivity, stroke rehabilitation assessment of movement and Fugl-Meyer lower extremity motor scale will also be conducted for subject characterization.

ELIGIBILITY:
Inclusion Criteria:

1. the diagnosis of first time unilateral stroke more than 6 months before
2. the ability to walk for at least 15 m without person assistance
3. apparent gait deficits upon visual inspection by a trained physical therapist or inability in community ambulation, i.e. walking speed < 0.8 m/s
4. resting blood pressure lower than 150/90 mmHg.

Exclusion Criteria:

1. older than 75 years
2. inability to follow the experimental instructions or procedures
3. any pain, inflammation, or other conditions that could affect walking
4. medically unstable.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
stride characteristics | 8 weeks
  Wearable movement sensors will be used to measure walking speed, stride length and time, and gait cycle.
  Ground reaction forces during walking. A force platform will be used to measure ground reaction forces and center of pressure.
Walking oxygen uptake | 8 weeks
  A Ultima Cordi 02 machine will be used to measure VO2 during 5-minute bouts of treadmill walking.
Balance | 8 weeks
  Berg Balance scale Minimum scale = 0 Maximum scale = 56 Higher scores indicate better functional balance.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No